CLINICAL TRIAL: NCT00385086
Title: Efficacy of TNF-alpha Inhibition in Sciatica With Post-operative Lumbar Spinal Fibrosis
Brief Title: Lumbar Spinal Fibrosis and TNF Alpha Inhibition
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P050312
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Post Operative Sciatica by Lumbar Spinal Fibrosis
Keywords: Sciatica; Pain; TNF-alpha; Discectomy; Fibrosis; Spine
MeSH Terms: conditions — Sciatica; Pain; Fibrosis | interventions — Tumor Necrosis Factor Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TNF-alpha blocker (Experimental): Treatment with TNF-alpha blocker
  Interventions: Drug: TNF blocker
- Placebo (Active Comparator): Treatment with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TNF blocker — Treatment with TNF-alpha blocker
  Arms: TNF-alpha blocker
Drug: Placebo — Treatment with placebo
  Arms: Placebo

SUMMARY:
TNF-alpha is the main cytokine implicated in the formation of lumbar spinal fibrosis. Inhibiting TNF-alpha could significantly decrease spinal fibrosis after lumbar discectomy.

DETAILED DESCRIPTION:
OBJECT:

Failed back surgery syndrome is still a challenging therapeutic problem. Clinical studies have demonstrated a significant association between lumbar spinal fibrosis after lumbar discectomy and the recurrence of radicular pain in 25% of cases. Forceful epidural infiltrations, radiotherapy, therapy with D-penicillamine or surgical procedures have had unfavourable results in terms of pain and cost. Magnetic resonance imaging reveals lumbar spinal fibrosis by a hyposignal in the T1 sequence and a hypersignal in T2 sequence around the spinal tissue. Tumor necrosis factor a (TNF-a) is the main cytokine implicated in the formation of tissue fibrosis. In animal models of fibrosis, TNF-a inhibition has been shown to prevent and treat tissue fibrosis.

HYPOTHESIS:

Inhibiting TNF-a could significantly decrease sciatica pain because of lumbar spinal fibrosis after lumbar discectomy by decreasing spinal fibrosis.

METHODS:

We propose a 2-year pilot prospective, randomized, double-blind, controlled study of TNF-a inhibitor (infliximab) in patients with sciatica as a result of postoperative lumbar spinal fibrosis. The infliximab group will receive one intravenous injection of 3 mg/kg infliximab. The control group will receive one physiological serum injection. Patients will be evaluated at day 0, 10, 30, 90, and 180. The main evaluation criterion will be sciatica pain as measured on a visual analog scale, with the objective of a 50% decrease in pain at day 10. This objective leads to a size of 20 patients per group. The other evaluation criteria will be clinical, functional, social, and professional. Patients will be recruited from the rehabilitation unit at Cochin teaching hospital.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old
* sciatica post discectomy
* Pain with VAS > 40 mm and impossibility to have his usual activity
* Surgical discectomy (less than 2 years and more than 6 months)
* Painless of more than one month and less than one year after the discectomy
* MRI with gadolinium injection of less than 6 months and done more than 6 months after the discectomy
* Presence of spinal fibrosis on MRI (hyposignal in T1 enhanced by gadolinium and hypersignal in T2)
* failure of epidural injection treatment
* absence of tuberculosis
* contraception for woman
* informed consent

Exclusion Criteria:

* Chronic psychiatric pathologies not treated
* Presence of conflict between nerve root and herniated disc or disc fragments or spinal stenosis
* severe cognitives troubles
* severe cardiac failure (class III or IV)
* Tuberculosis (active or latent), severe infections
* Cancers
* Allergy reactions to the drug studied
* Difficulties to understand french
* Patients enrolled in another clinical trial in the past three months
* pregnancy, breastfeeding or no contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-02; Primary Completion 2012-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Sciatica pain | 10 days after treatment
  Visual analogue scale of lumbar pain

SECONDARY OUTCOMES:
Functional assessments | At 10, 30, 90, 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Francois Rannou, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Cochin, Paris, Paris, France

REFERENCES:
- [Derived] Nguyen C, Palazzo C, Grabar S, Feydy A, Sanchez K, Zee N, Quinquis L, Ben Boutieb M, Revel M, Lefevre-Colau MM, Poiraudeau S, Rannou F. Tumor necrosis factor-alpha blockade in recurrent and disabling chronic sciatica associated with post-operative peridural lumbar fibrosis: results of a double-blind, placebo randomized controlled study. Arthritis Res Ther. 2015 Nov 19;17:330. doi: 10.1186/s13075-015-0838-4. PMID 26596627